CLINICAL TRIAL: NCT02123914
Title: Effects of Chronic Exercise Training and Vitamin C Supplementation on Physiological Changes and Symptoms in Allergic Rhinitis Patients
Brief Title: The Effect of Exercises on Physiological Changes and Clinical Symptoms in Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr.Daroonwan Suksom, Faculty of Sports Science, Chulalongkorn University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: SPSC-2
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Allergic Rhinitis
Keywords: Exercise training; Allergic rhinitis; Vitamin C; Cytokine; Rhinitis symptoms
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Exercise; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise with Vit. C & Aerobic exercise (Experimental)
  Interventions: Other: Aerobic exercise with Vit. C; Other: Aerobic exercise
- exercise without vit. c supplement & no exercise (Active Comparator)
  Interventions: Other: Aerobic exercise with Vit. C; Other: No exercise

INTERVENTIONS:
Other: Aerobic exercise with Vit. C — walking - running on a treadmill at intensity of 65-70% HRR for 30 minutes per session three times a week combined with taking vitamin C supplemented daily with an oral dose of 2,000 mg 2 times/day for 8 weeks.
  Nasal challenge with house dust mites with the evaluation of cytokines in nasal lavage fluid,
  Nasal peak flow measurement,
  Nasal blood flow measurement,
  Exercise training regimen including VO2max measurment at baseline and at the end of the experiment.
Other: Aerobic exercise — walking - running on a treadmill at intensity of 65-70% HRR for 30 minutes per session three times a week for 8 weeks.
  Nasal challenge with house dust mites with the evaluation of cytokines in nasal lavage fluid,
  Nasal peak flow measurement,
  Nasal blood flow measurement,
  Exercise training regimen including VO2max measurment at baseline and at the end of the experiment.
  Arms: Aerobic exercise with Vit. C & Aerobic exercise
Other: No exercise — Sedentary control.
  Nasal challenge with house dust mites with the evaluation of cytokines in nasal lavage fluid,
  Nasal peak flow measurement,
  Nasal blood flow measurement,
  Exercise training regimen including VO2max measurment at baseline and at the end of the experiment.
  Arms: exercise without vit. c supplement & no exercise

SUMMARY:
1. Moderate exercise training decrease cytokine response and rhinitis symptoms in patients with allergic rhinitis
2. Moderate exercise training combined with vitamin C supplementation decrease cytokine response and rhinitis symptoms in patients with allergic rhinitis
3. Moderate exercise training combined with vitamin C supplementation has more beneficial effects than moderate exercise training alone for decreasing cytokine response and rhinitis symptoms in patients with allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria included patients with allergic rhinitis who had a clinical history of persistent rhinitis, and had positive skin prick test (wheal diameter ≥ 3 mm) to house dust mite (D. pteronyssinus).

Exclusion Criteria:

Subjects with known asthma, chronic rhinosinusitis, hypertension or cardiovascular diseases were excluded.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in rhinitis symptoms | Baseline, week 8
  Nasal symptoms will be assessed using a rhinitis symptom score questionnaire. The subjects will be asked to score symptoms of persistent allergic rhinitis; nasal congestion, itching, sneezing, and rhinorrhea before and after each exercise protocol. The score ranged from 0 to 3 points (0 = none, 1 = mild, 2 = moderate, 3 = severe).
Changes from baseline in cytokine | baseline, week 8
  The cytokines IL-2, IL-4, and IL-13 in blood and nasal secretion will be determined by using the flow cytometry technique (Scavuzzo MC. et al., 2003). Data will be acquired using a flow cytometer (BD FACSCalibur Flow Cytometer, USA) and analyzed by FlowcytomixTM Pro software (eBioscience, USA.).

SECONDARY OUTCOMES:
Changes from baseline in pulmonary function | Baseline, Week 8
  Pulmonary function (FVC and FEV1) will be conducted on all subjects using a calibrated computerized pneumotachograph spirometer (Spirotouch; Burdick, Inc., Deerfield, Wisconsin USA.) according to American Thoracic Society (ATS) recommendations (Laszlo G., 2006).
Changes from baseline in cardiorespiratory fitness (VO2max) | Baseline, Week 8
  VO2max will be performed using bruce treadmill protocol. Subjects will be asked to run on a treadmill (Landice, USA) in which the grade and intensity will be increased every 3 minutes until exhaustion.
Changes from baseline in nasal blood flow | Baseline, week 8
  Nasal mucosa blood flow will be measured by laser doppler flowmetry (DRT4 moor instrument, UK.). A side delivery endoscopic probe with flexible nylon sleeve with a diameter of 1.34 mm was placed on the anterior surface of the nose. The nasal blood flow values before and after exercise in each protocol will be then measured.
Changes from baseline in peak nasal inspiratory flow | Baseline, Week 8
  Peak nasal inspiratory flow (PNIF) will be measured using a peak nasal inspiratory flow meter (Clement Clark International model IN-CHECK ORAL, UK.) attached to an anesthesia mask. During the procedure, the subjects placed a mask over the nose and mouth and inspired forcefully through the nose, with lips tightly closed. PNIF will be measured before and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Daroonwan Suksom, Ph.D., Principal Investigator — Faculty of Sports Science, Chulalongkorn University
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Patumwan, Bangkok, Thailand

REFERENCES:
- [Background] Klaewsongkram J, Ruxrungtham K, Wannakrairot P, Ruangvejvorachai P, Phanupak P. Eosinophil count in nasal mucosa is more suitable than the number of ICAM-1-positive nasal epithelial cells to evaluate the severity of house dust mite-sensitive allergic rhinitis: a clinical correlation study. Int Arch Allergy Immunol. 2003 Sep;132(1):68-75. doi: 10.1159/000073266. PMID 14555860